CLINICAL TRIAL: NCT04506723
Title: Comparison of the Morphological Picture of the Renal Parenchyma With the Results of Mathematical Analysis of Intrarenal Transport of Contrast Medium in Computed Tomography in Patients With Urolithiasis
Brief Title: Comparison of Morphological and Radiological Data in Patients With Urolithiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy Director for Research, I.M. Sechenov First Moscow State Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Stone-CL-01
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with urolithiasis (Experimental): Patients with confirmed urolithiasis who is assigned to PCNL.
  Interventions: Procedure: Percutaneous Nephrolithotomy
- Patients without urolithiasis (Active Comparator): Patients with renal tumor without urolithiasis in history who is assigned to partial or radical nephrectomy due to renal tumor.
  Interventions: Procedure: Partial nephrectomy; Procedure: Radical nephrectomy

INTERVENTIONS:
Procedure: Percutaneous Nephrolithotomy — PCNL will be carried out in accordance with the standards and capabilities of the medical center. After the procedure pathomorphological data of the renal parenchyma will be assessed
  Arms: Patients with urolithiasis
Procedure: Partial nephrectomy — Partial nephrectomy will be carried out in accordance with the standards and capabilities of the medical center. After the procedure pathomorphological data of the renal parenchyma will be assessed
  Arms: Patients without urolithiasis
Procedure: Radical nephrectomy — Nephrectomy will be carried out in accordance with the standards and capabilities of the medical center. After the procedure pathomorphological data of the renal parenchyma will be assessed
  Arms: Patients without urolithiasis

SUMMARY:
The aim of the study was to compare the ultrastructural changes in the renal parenchyma with the results of postprocessing CT analysis with contrast enhancement in patients with urolithiasis.

ELIGIBILITY:
Inclusion Criteria for experimental group:

1. Men and women >18 years and <45 years old;
2. Established diagnosis of urolithiasis that does not interfere with the processes of urodynamics (there is no expansion of the overlying urinary tract);
3. Planned surgery - percutaneous nephrolithotripsy;
4. Stone size up to 20 mm., Patients with multiple small two-sided stones;
5. Patients with CT of the kidneys with contrast enhancement performed according to the required protocol.

Exclusion Criteria for experimental group:

1. Age < 18 years old or ASA> 3;
2. With single kidney;
3. Patients with coral stones;
4. The presence of concomitant systemic pathology (DM, AH), as well as kidney disease (glomerulonephritis), which can change the state of the renal parenchyma;
5. A history of injuries and surgical interventions on the kidneys, urinary tract, renal vessels;
6. Taking nephrotropic drugs;
7. Systemic intake of nephrotoxic drugs;
8. Severe general somatic condition, making the operation impossible;
9. Pregnancy.

Inclusion Criteria for control group:

1. Men and women >18 years and <45 years old;
2. Absence of urolithiasis in the patient's anamnesis and in his family history;
3. Renal tumors which have undergone partial nephrectomy or nephrectomy;
4. Patients with CT renal data with contrast enhancement, performed according to the required protocol.

Exclusion Criteria for control group:

1. Urolithiasis in anamnesis;
2. A history of trauma and surgical interventions on the kidneys, urinary tract, renal vessels;
3. Intercurrent background;
4. Non-informative biopsy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the features of interrenal transport of contrast agent and the structural state of the renal tissue | 1 month
  The data of 3D analysis of CT of the kidneys in patients with urolithiasis

SECONDARY OUTCOMES:
To assess the features of the morphological structure of glomeruli, tubules, perivascular and interstitial spaces of renal tissue in patients with urolithiasis | 2 weeks
  The assessment will be based on intraoperative biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Enikeev, M.D., Ph.D., Study Director — Sechenov University; Dmitry Fiev, M.D., Ph.D., Principal Investigator — Sechenov University
Locations (1):
- Institute for Urology and Reproductive Health, Sechenov University., Moscow, Russia

IPD SHARING:
Plan to Share IPD: No